CLINICAL TRIAL: NCT03386708
Title: A Clinical Research on the Safety/Efficacy of Human Umbilical Cord Mesenchymal Stem Cell (19#iSCLife®-CSD) Therapy for Patients With Healing Poor After Uterus Injury
Brief Title: hUC Mesenchymal Stem Cells (19#iSCLife®-CSD) Therapy for Patients With Healing Poor After Uterus Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sclnow Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLnow-XY-01
Record Dates: First submitted 2017-12-12; First posted 2017-12-29 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2021-09

CONDITIONS: Uterus; Injury
Keywords: Healing Poor After Uterus Injury, Mesenchymal Stem Cell
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hUC-MSC intrauterine injection group (Experimental): Human umbilical cord mesenchymal stem cells (hUC-MSC) (SCLnow 19#)
  Interventions: Procedure: intrauterine injection; Biological: human umbilical cord mesenchymal stem cell

INTERVENTIONS:
Procedure: intrauterine injection — intrauterine injection with umbilical cord mesenchymal stem cell (SCLnow 19#); one time/one menstrual cycle, total 2 times
Biological: human umbilical cord mesenchymal stem cell — 2 * 10^7 cells (2ml)

SUMMARY:
The purpose of this study is verify the efficacy and safety of Human Umbilical Cord Mesenchymal Stem Cells (UC-MSC) therapy for patients with Healing Poor after Uterus Injury, and exploring the possible mechanisms of umbilical cord mesenchymal stem cell therapy in Healing Poor After Uterus Injury disease

DETAILED DESCRIPTION:
This is a random, open label, and self-control experiment. 10 patients are selected and sign consent forms, then divided into one group. Doctors collect the basic information of patient (including age,height, mental condition, vital sign, history of disease, pharmaco-history, and so on.), evaluate the symptom of healing Poor after Uterus Injury (Menstrual conditions, Visual analogue scale, pregnancies).

All patients receive laboratory and image examination as baseline. Then, cell treatment will be given based on the clinical protocol. Doctors have follow-up visit on 3 and 6 month after treatment, and do efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Female, with BMI 18-24 kg/m^2
* Meet the clinical standard of Healing Poor After Uterus Injury
* Non smoker
* Do not accept stem cells treatment in 6 months
* Participants or their family members sign the consent form of this study

Exclusion Criteria:

* Pregnant or breast feeding women
* Age <18 or >40
* Refuse to sign the consent form
* Patients with underlying risk of medical disease history: history of diabetes, serious cardiovascular disease, severe infection, alimentary tract hemorrhage, etc.
* Serum with HIV, syphilis antibody positive
* Severe mental disease, cognitive disorder patients
* Other severe system or organ organic disease
* Participate other clinical experiments in 3 months
* Ovarian and pituitary dysfunction diseases
* With some other conditions that doctor propose not to participate

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Intrauterine adhesion patients efficacy evaluation | 12 months
  Evaluate the efficacy by calculating the thickness of endometrium, the equation is, Efficacy = (thickness of endometrium after treatment - thickness of endometrium before treatment)/thickness of endometrium before treatment * 100%
  Classified the efficacy in 4 grade as follow, A. Recovery, efficacy 86% - 100%; B. Obvious improve, efficacy 46% - 85%; C. Improve, efficacy 16% -45%; D. Invalid, efficacy < 16% Grade A, B, and C is proposed to be effective.

SECONDARY OUTCOMES:
Incision lacuna and incision diverticulum patients efficacy evaluation | 12 months
  Evaluate the efficacy by calculating the 50% or more reduction, the equation is, Efficacy = (Area of lacuna and diverticulum after treatment - Area of lacuna and diverticulum after treatment before treatment)/Area of lacuna and diverticulum before treatment * 100%.
  Classified the efficacy in 4 grade as follow, A. Recovery, efficacy 86% - 100%; B. Obvious improve, efficacy 46% - 85%; C. Improve, efficacy 16% -45%; D. Invalid, efficacy < 16% Grade A, B, and C is proposed to be effective.
Ultrasound of uterus evaluation | 12 months
  Ultrasound of uterus. Compare with the baseline images, evaluate the changes/improvement after cell treatment.
Hysteroscopy evaluation | 12 months
  Do hysteroscopy examination, compare with the baseline images, evaluate the change/improvement after cell treatment.
Pain score | 12 months
  Measure the pain score of patients by Visual Analog Score (VAS) for pain

CONTACTS AND LOCATIONS:
Overall Officials: Weishe Zhang, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

REFERENCES:
- [Derived] Huang J, Li Q, Yuan X, Liu Q, Zhang W, Li P. Intrauterine infusion of clinically graded human umbilical cord-derived mesenchymal stem cells for the treatment of poor healing after uterine injury: a phase I clinical trial. Stem Cell Res Ther. 2022 Mar 3;13(1):85. doi: 10.1186/s13287-022-02756-9. PMID 35241151